CLINICAL TRIAL: NCT00977626
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of Oral AZD2423 Solution After Multiple Ascending Doses in Young and Elderly Healthy Volunteers
Brief Title: Study to Investigate Safety, Tolerability and Pharmacokinetics of AZD2423 Multiple Doses in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D2600C00002
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Healthy; Pharmacokinetics; Healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 AZD2423 or Placebo (Experimental): AZD2423 or Placebo Oral Solution, multiple dosing during 10-14 days
  Interventions: Drug: Part 1 - AZD2423 or Placebo
- Part 2 - AZD2423 (Experimental): AZD2423 Oral solution, multiple dosing
  Interventions: Drug: Part 2 - AZD2423
- Part 3 - AZD2423 (Experimental): AZD2423 Oral solution single dosing or AZD2423 Oral solution, single dosing - With Food or AZD2423 Oral solution, single dosing - Fasting Condition.
  Interventions: Drug: Part 3 - AZD2423

INTERVENTIONS:
Drug: Part 1 - AZD2423 or Placebo — AZD2423 Oral Solution, multiple dosing during 10-14 days or Placebo Oral Solution, multiple dosing during 10-14 days
  Arms: Part 1 AZD2423 or Placebo
Drug: Part 2 - AZD2423 — AZD2423 Oral solution, multiple dosing
  Arms: Part 2 - AZD2423
Drug: Part 3 - AZD2423 — AZD2423 Oral solution, single dosing or AZD2423 Oral solution, single dosing - With Food or AZD2423 Oral solution, single dosing - Fasting Condition.
  Arms: Part 3 - AZD2423

SUMMARY:
Three-part study investigating the safety and tolerability of AZD2423 multiple doses in 98 healthy volunteers: Part 1 80 young and elderly subjects in a parallel, double blind, randomised study. Part 2 - 6 subjects in an open, non-randomised study. Part 3 - 12 subjects in a three-way cross over, open label, partially randomised study.

Part 1 has 2 Arms, AZD2423 or Placebo, Multiple dosing during 10-14 days . Part 2 has 1 Arm AZD2423 Multiple dosing and Part 3 has 3 Arms AZD2423 single dosing or AZD2423 single dosing with food or AZD2423 single dosing, Fasting Condition

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Healthy male and non-fertile female subjects aged ≥20 to ≤55 years inclusive and healthy male and female subjects aged ≥65 to ≤80 years inclusive with suitable veins for cannulation or repeated venepuncture.
* Have a body mass index (BMI) between ≥18 and ≤30 kg/m2, as calculated by the investigator, and weigh at least 50 kg and no more than 100 kg.
* Clinically normal physical findings including supine blood pressure, pulse rate, ECG, and laboratory assessments in relation to age, as judged by the investigator. In addition, normal ophthalmoscopy is required for the CSF panel subjects (Part 2).

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study,or influence the results or the subject's ability to participate in the study
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
* Any clinically significant illness/infection or medical/surgical procedure or trauma, as judged by the Principal Investigator, within 3 months of the first administration of investigational product.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Investigate the safety and tolerability of AZD2423 in young and elderly subjects following multiple ascending doses at steady state and, if possible, estimate the maximum tolerated dose if within the predefined exposure limits (Part 1 and 2 only). | Part 1:Safety samples taken frequently throughout the study at screening, d-1 and from days 2-16 and at the follow up visit. Part 2: Safety samples taken frequently throughout the study at screening, d-1 and from days 1-9 and at follow up visit.

SECONDARY OUTCOMES:
Characterize multiple dose PK of AZD2423 and assess time required to reach steady state, degree of accumulation and time dependency of PK (Part 1 and Part 2 only). Characterize single and multiple dose PK of AZD2423 in elderly subjects (Part 1 only) | Part 1: PK will be taken days 1-14 inclusive and at follow-up, with a full PK day on Day 1 and 14. Part 2: PK samples taken on days 1-9 and at follow up visit. Day 1 and 8 is a full PK day.
To investigate concentration of AZD2423 in cerebrospinal fluid (CSF) (Part 2 only). | Part 2: CSF Samples will be taken on day 8 at 4 and 24 hours post dose.
Investigate the PK of tablet formulation compared to oral solution, effect of food compared to fasting, and investigate the safety and tolerability of oral solution and tablet formulation of AZD2423 in young subjects after admin. of single dose (Part 3) | Safety samples taken frequently throughout the study at screening, d-1 and from days 2+3 7-10, 14, 16+17 and at the follow up visit. PK samples will be taken on days 1-4, 8-11, 15-18 and at the follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Muna Albayaty, Principal Investigator — PAREXEL Early Phase Clinical Uniit, London; Richard Malamut, Study Director — AstraZeneca R&D
Locations (1):
- Research Site, Harrow, United Kingdom